CLINICAL TRIAL: NCT02796976
Title: Exercise, Arterial Cross-Talk Modulation and Inflammation in an Ageing Population (ExAMIN AGE)
Brief Title: Exercise, Arterial Cross-Talk Modulation and Inflammation in an Ageing Population
Acronym: ExAMIN AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Basel Institute of Clinical Epidemiology (BICE) (Other)
Responsible Party: Principal Investigator, Henner Hanssen, Prof. Dr. med. Henner Hanssen, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ-2015-351
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Cardiovascular Disease; Obesity; Atherosclerosis; Heart; Disease, Activity
Keywords: arterial stiffness; retinal vessels; physical activity; ageing
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Atherosclerosis; Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- healthy older active (No Intervention): only cross-sectional
- healthy older sedentary (No Intervention): only cross-sectional
- older sedentary at risk (Active Comparator): cross-sectional and training or control condition
  Interventions: Other: Training or control condition

INTERVENTIONS:
Other: Training or control condition — Participants get a 12 week high intensity and walking-based interval training which is adapted to their individual physical fitness level or a general recommendation on physical activity according to European Guidelines.
  Arms: older sedentary at risk

SUMMARY:
The aims of the study are twofold. In the cross-sectional approach (Part I), the study will be conducted in an older population to assess the association of physical fitness on different parts of the human vascular bed. In the interventional approach (Part II), it aims to investigate whether and to what extent advanced vascular ageing (AVA) in older subjects with increased cardiovascular risk can be reversed by regular walking- based high intensity interval training.

DETAILED DESCRIPTION:
In the cross-sectional part the investigators analyze physical fitness, vascular health and further outcomes in a healthy older active, a healthy older sedentary and a obese sedentary group with increased cardiovascular risk. The investigators will analyze large and small artery function, physical fitness and activity as well as inflammatory parameters in these three groups. Here the investigators will investigate the influence of physical activity and inflammatory parameters on the vascular health in different beds.

In the intervention part the older sedentary group with increasing cardiovascular risk (OSR) will be randomized in a control and an intervention group. The intervention group will get a high intensity interval training which is walking based and individual adjusted. The control group will get general lifestyle recommendations. After 12 weeks of training OSR group will be tasted again. The aim of the second part is to assess the effect of high intensity interval training on vascular health and inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 50-79 years
* Active lifestyle: > 9 MET/week (> 3hours moderate walking/week); 18.5≤ BMI ≤ 29.9 kg/m2
* Sedentary lifestyle: ≤ 3 MET/week (≤ 1 hour moderate walking/week); 18.5≤ BMI ≤ 29.9 kg/m2
* Sedentary men and women aged 50-79 years with increased cardiovascular risk are allowed to have ≥ one additional cardiovascular risk factor

Exclusion Criteria:

* History of cardiovascular, pulmonary or chronic inflammatory disease
* blood pressure ≥ 140/90 mmHg during 24h monitoring
* current or past smoker (in healthy group)
* macular degeneration or glaucoma
* compromising orthopaedic problems

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change of pulse wave velocity (m/s) | Change from baseline pulse wave velocity at 12 weeks
  Measured at local, central and peripheral site

SECONDARY OUTCOMES:
Change of augmentation index (AIx@75) in % | Change from baseline augmentation index at 12 weeks
  AIx and AIx@75 will be measured by using the gold standard device for single measurements (SphygmoCor®)
Change of arteriolar to venular diameter ratio (AVR) in µm | Change from baseline AVR at 12 weeks
  Dynamic and static retinal vessel analyzes will be investigated
Change of physical activity in METs per week | Change from baseline physical activity at 12 weeks
  The Freiburger Questionnaire of physical activity and inactivity and an accelerometer for seven days will be used to measure physical activity.
Change of physical fitness in VO2max | Change from baseline VO2max at 12 weeks
  An individual treadmill ramp test will be used to investigate peak oxygen consumption and maximal heart rate.

OTHER OUTCOMES:
Change of diastolic function parameters (E/A; E/E') | Change from baseline parameters at 12 weeks
  Echocardiography
Change of autonomic function in heart rate variability (HRV) in beats per minute (bpm) | Change from baseline HRV at 12 weeks
  12-lead ECG monitoring
Change of serum biomarkers (hs-CRP, IL-6, IL-10, TNF-α) | Change from baseline serum biomarkers at 12 weeks
  Blood sampling
Change of cognitive Function | Change from baseline cognitive function at 12 weeks
  Executive function test battery

CONTACTS AND LOCATIONS:
Locations (1):
- Bereich Sport- und Bewegungsmedizin, Abteilung Präventive Sportmedizin & Systemphysiologie, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanssen H, Nussbaumer M, Moor C, Cordes M, Schindler C, Schmidt-Trucksass A. Acute effects of interval versus continuous endurance training on pulse wave reflection in healthy young men. Atherosclerosis. 2015 Feb;238(2):399-406. doi: 10.1016/j.atherosclerosis.2014.12.038. Epub 2014 Dec 23. PMID 25558034
- [Background] Nussbaumer M, Donath L, Fischer M, Schafer J, Faude O, Zahner L, Schmidt-Trucksass A, Hanssen H. Effects of acute bouts of endurance exercise on retinal vessel diameters are age and intensity dependent. Age (Dordr). 2014 Jun;36(3):9650. doi: 10.1007/s11357-014-9650-3. Epub 2014 Apr 12. PMID 24728623
- [Background] Hanssen H, Nickel T, Drexel V, Hertel G, Emslander I, Sisic Z, Lorang D, Schuster T, Kotliar KE, Pressler A, Schmidt-Trucksass A, Weis M, Halle M. Exercise-induced alterations of retinal vessel diameters and cardiovascular risk reduction in obesity. Atherosclerosis. 2011 Jun;216(2):433-9. doi: 10.1016/j.atherosclerosis.2011.02.009. Epub 2011 Feb 17. PMID 21392768
- [Derived] Streese L, Demougin P, Iborra P, Kanitz A, Deiseroth A, Kropfl JM, Schmidt-Trucksass A, Zavolan M, Hanssen H. Untargeted sequencing of circulating microRNAs in a healthy and diseased older population. Sci Rep. 2022 Feb 22;12(1):2991. doi: 10.1038/s41598-022-06956-4. PMID 35194110
- [Derived] Deiseroth A, Streese L, Kochli S, Wust RS, Infanger D, Schmidt-Trucksass A, Hanssen H. Exercise and Arterial Stiffness in the Elderly: A Combined Cross-Sectional and Randomized Controlled Trial (EXAMIN AGE). Front Physiol. 2019 Sep 4;10:1119. doi: 10.3389/fphys.2019.01119. eCollection 2019. PMID 31551805
- [Derived] Streese L, Kotliar K, Deiseroth A, Infanger D, Vilser W, Hanssen H. Retinal Endothelial Function, Physical Fitness and Cardiovascular Risk: A Diagnostic Challenge. Front Physiol. 2019 Jul 5;10:831. doi: 10.3389/fphys.2019.00831. eCollection 2019. PMID 31333489
- [Derived] Streese L, Khan AW, Deiseroth A, Hussain S, Suades R, Tiaden A, Kyburz D, Cosentino F, Hanssen H. High-intensity interval training modulates retinal microvascular phenotype and DNA methylation of p66Shc gene: a randomized controlled trial (EXAMIN AGE). Eur Heart J. 2020 Apr 14;41(15):1514-1519. doi: 10.1093/eurheartj/ehz196. PMID 31323685